CLINICAL TRIAL: NCT01074255
Title: Re-examination Study For General Drug Use to Assess the Safety and Efficacy Profile of EMEND in Usual Practice
Brief Title: Re-examination Study of EMEND (Aprepitant) (MK-0869-184)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0869-184; MK-0869-184 (Other: protocol number)
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2012-10-05 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: Nausea; Vomiting; Chemotherapy; Post-chemotherapy
MeSH Terms: conditions — Vomiting; Nausea | interventions — Aprepitant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Korean Participants Treated With EMEND (aprepitant): Participants receiving EMEND on Treatment Days 1, 2, and 3 concomitantly with a corticosteroid and a 5-hydroxytryptamine 3 (5-HT3) antagonist.
  Interventions: Drug: EMEND

INTERVENTIONS:
Drug: EMEND — EMEND (Aprepitant,125 mg oral capsules) is administered 1 hour prior to chemotherapy on treatment Day 1. EMEND (80 mg) is administered on the morning of Days 2 and 3. EMEND is concomitantly administered with a regimen of a corticosteroid and a 5-HT3 antagonist.
  Other Names: Aprepitant; MK-0869

SUMMARY:
This survey is conducted for preparing application materials for re-examination under the Pharmaceutical Affairs Laws and its Enforcement Regulation. Its aim is to reconfirm the clinical usefulness of EMEMD (aprepitant) through collecting the safety information according to the Re-examination Regulation for New Drugs.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are treated with EMEND for the first time as per the EMEND label

Exclusion Criteria:

* Contraindication to EMEND

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean patients treated with EMEND in usual practice.
Sampling Method: Probability Sample
Enrollment: 3546 (Actual)
Dates: Start 2007-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: South Korean hospitals provided 3,546 participant's case report forms, 9/18/2006-1/22/2012. 407 participants were excluded: 201 violated dosage/administration, 173 lost to follow-up, 15 duplicated participants, 10 assessed before the contracted date, 3 previously received EMEND, 3 violated inclusion/exclusion criteria, and 2 didn't receive EMEND.
Groups:
- Korean Participants Treated With EMEND (Aprepitant): EMEND (125 mg oral capsules) is administered 1 hour prior to chemotherapy on Treatment Day 1. EMEND (80 mg) is administered on the morning of Days 2 and 3. EMEND is concomitantly administered with a regimen of a corticosteroid and a 5-HT3 antagonist.
Period: Overall Study
Arm/Group | Korean Participants Treated With EMEND (Aprepitant)
Started | 3141
Treated | 3139
Completed | 3139
Not Completed | 2
Not completed — Did not receive EMEND | 2

BASELINE CHARACTERISTICS:
Arm/Group | Korean Participants Treated With EMEND (Aprepitant)
Number analyzed (Participants) | 3139
Age, Customized [Number; unit: Participants]
  <40 years | 296
  40 to 49 years | 635
  50 to 59 years | 898
  60 to 69 years | 957
  ≥70 years | 353
Sex/Gender, Customized [Number; unit: Participants]
  Male | 1729
  Female | 1410

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment of Participants' Response to Therapy With EMEND (Aprepitant) for the Prevention of Acute and Delayed Nausea Following Chemotherapy
Description: The investigators assessed a participant's response to therapy with EMEND to prevent acute and delayed nausea and vomiting associated with initial and repeat courses of chemotherapy when used concomitantly with other antiemetics. The response categories were: excellent (best possible anticipated response, considering the severity and stage of disease), good (good response, but less than the best possible anticipated response), fair (definite response, but could be better), poor (minimal response, unacceptable), or none (no response, absence of drug effect).
Time Frame: Up to 14 days following the cessation of treatment
Population: The Efficacy Evaluable Population consisted of participants treated with EMEND for 3 days and assessed by an investigator for efficacy. Participants were excluded from efficacy analysis for having a EMEND administration period less than 3 days (143 participants) or unavailability of final efficacy evaluation (1 participant).
Measure: Number; unit: participants
Arm/Group | Participants Treated With EMEND
Number analyzed (Participants) | 2995
participants
  Excellent | 438
  Good | 2056
  Fair | 446
  Poor | 52
  None | 3

ADVERSE EVENTS:
Time Frame: Up to 14 days following the cessation of treatment
Description: Participants who completed more than one follow up visit were included in the cases for safety evaluation.
Groups:
- Participants in the Safety Analysis: Participants included in the Safety Analysis
Arm/Group | Participants in the Safety Analysis
Serious Adverse Events (participants affected / at risk) | 89/3139
Other Adverse Events (participants affected / at risk) | 399/3139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants in the Safety Analysis (N=3139)
Nausea (Gastrointestinal disorders) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 17 (17)
Mucosal inflammation (General disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 22 (22)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 14 (14)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
White blood cell count decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 2 (2)
Pneumonia (Infections and infestations) | 7 (7)
Oral candidiasis (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 3 (3)
Septic shock (Infections and infestations) | 4 (4)
Nephropathy toxic (Renal and urinary disorders) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Infarction (Vascular disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Gastritis atrophic (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 4 (4)
Multi-organ failure (General disorders) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants in the Safety Analysis (N=3139)
Nausea (Gastrointestinal disorders) | 281 (285)
Decreased Appetite (Metabolism and nutrition disorders) | 195 (195)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator intends to publish trial results in an academic journal, prior consent of the sponsor must be obtained.